CLINICAL TRIAL: NCT04219631
Title: Results of Regulated Expiratory Breathing Method During Childbirth Process
Brief Title: Regulated Expiratory Breathing Method During Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Kaouther Dimassi, associate professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Winner flow-URO- MG Mongi Slim
Record Dates: First submitted 2019-12-19; First posted 2020-01-07 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Childbirth
Keywords: delivery; cesarean; expiration; exercise; labor
MeSH Terms: conditions — Death; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WINNER- FLOW-URO-MG GROUP (Experimental): After admission to the delivery room, all women assigned to WF + group will have an interview with one of the midwifes responsible for the study. The latter will explain the use of the WINNER FLOW®-URO MG® device which is the expiration mouthpiece used during breathing exercises to ensure a constant ventilatory flowrate. Then, WF+ patients will use the expiratory mouthpiece device during all their childbirth process.
  Interventions: Device: expiration mouthpiece used during breathing exercises to ensure a constant ventilatory flowrate.
- NO WINNER-FLOW-URO-MG GROUP (No Intervention): Women enrolled in WF- group will be managed classically during their child birth process regardless to the study participation.

INTERVENTIONS:
Device: expiration mouthpiece used during breathing exercises to ensure a constant ventilatory flowrate. — women enrolled in WINNER-FLOW-URO-MG group will freely use the expiratory mouthpiece device during all their childbirth process.
  Arms: WINNER- FLOW-URO-MG GROUP

SUMMARY:
The factors affecting the rate of primary caesarean section births are complex, and identifying interventions to reduce this rate is challenging. Effective interventions targeting at women are mainly represented by Childbirth training workshops, psychoeducation and psychosocial couple-based programs. Considering non medical interventions targeting mothers, the pattern of breathing during labor that can help for vaginal delivery is a controversial topic. There are no data to support a policy of directed maternal breathing or pushing during vaginal delivery.

The abdomino-perineal concept was originally a postpartum rehabilitation technique. Currently, applications are increasing. During labor, expiration channeled by a flow regulator device offers support to women enduring the pain of uterine contractions. During the second stage, the expiratory regulated pushing allows a long, efficient and very intuitive push.

The use of this regulated expiratory breathing method was introduced in the study unit in January 2018. Despite a positive experience both reported by women and midwives, investigators have so far only subjective feedback without objective measurable clinical impact.

As a result, investigators are conducting this scientific study whose main objective is:

- To Evaluate the impact of a regulated expiratory breathing method on childbirth process .

DETAILED DESCRIPTION:
Rates of cesarean delivery continue to rise worldwide, with recent (2016) reported rates of 24.5% in Western Europe, 32% in North America, and 41% in South America.

Primary cesarean deliveries account for more than half of all cesarean deliveries, and the most common indication for repeat cesarean delivery is previous cesarean delivery.

Consequently, the reduction in primary cesarean delivery rate represents a meaningful objective.

The factors affecting the rate of primary caesarean section births are complex, and identifying interventions to reduce this rate is challenging. Effective interventions targeting at women are mainly represented by Childbirth training workshops, psychoeducation and psychosocial couple-based programs. Considering non medical interventions targeting mothers, the pattern of breathing during labor that can help for vaginal delivery is a controversial topic. There are no data to support a policy of directed maternal breathing or pushing during vaginal delivery.

The abdomino-perineal concept was originally a postpartum rehabilitation technique. Currently, applications are increasing. Currently, applications are increasing. During labor, expiration channeled by a flow regulator device offers support to women enduring the pain of uterine contractions. During the second stage, the expiratory regulated pushing allows a long, efficient and very intuitive push.

The use of this regulated expiratory breathing method was introduced in the study unit in January 2018. Despite a positive experience both reported by women and midwives, we investigators have so far only subjective feedback without objective measurable clinical impact.

As a result, investigators are conducting this scientific study whose main objective is:

- To Evaluate the impact of a regulated expiratory breathing method on childbirth process .

ELIGIBILITY:
Inclusion Criteria:

* Primiparae
* Singleton pregnancy
* Gestational age ≥ 37 SA
* Fetus in cephalic presentation
* Fetus with a normal weight for a the gestational age
* Spontaneous onset of labor
* Early stage of labor (with cervical dilatation under 3 cm)
* No previous Childbirth training workshops

Exclusion Criteria:

* Parity of at least 2
* Multiple pregnancy
* Intra uterine fetal demise
* Previous uterine scar
* Fetus in Breach presentation
* Non Vertex cephalic presentation
* Narrowed pelvic bone diameters
* A contraindication to vaginal delivery (placenta previa , fibroma previa, …)
* Previous participation to childbirth training workshops
* Women in an advanced stage of labor with a cervical dilation upon admission over 3 cm
* Women requiring epidural anesthesia
* Refusal of participation

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
cesarean delivery rate | through study completion, an average of 1 year
  percentage of cesarean delivery in each group

SECONDARY OUTCOMES:
Duration of first stage of labor | up to 10 hours . In deed , For each recruited patient this outcome will be measured in minutes between onset of labor and achievement of complete cervical dilation
  For each recruited patient this outcome will be measured in minutes between onset of labor and achievement of complete cervical dilation
Duration of the second stage of labor | up to one hour . In deed, investigators will measure for each included patient the time ( minutes ) elapsed from complete cervical dilation and newborn delivery
  For each included patient investigators will measure in minutes the time elapsed from complete cervical dilation and newborn delivery
duration of placental delivery | up to 20 minutes .Investigators will measure for each included patient the time in minutes elapsed between newborn delivery and placental expulsion.
  Investigators will measure for each included patient the time in minutes elapsed between newborn delivery and placental expulsion.
Rate of Spontaneous vaginal birth | through study completion, an average of 1 year
  percentage of natural vaginal birth in each group
Rate of Instrumental vaginal birth | through study completion, an average of 1 year
  percentage of use of forceps in case of vaginal birth
Episiotomy rate | through study completion, an average of 1 year
  percentage of episiotomy in case of vaginal delivery in each group
rate of Intra-partum Fetal compromise | through study completion, an average of 1 year
  percentage of fetal heart rate observed during labor and delivery in each group
Pain scores during labor and delivery | four times: up yo one hour, up to four hours, up to 8 hours , up to 10 hours
  pain assessment will use Visual Analogue Scale for Pain (VAS Pain) intensity ( The pain VAS is a single-item scale.For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale] )
  During childbirth process, pain assessment will be repeated four times:
  First assessment during early first stage of labor with a cervix dilation less than 3 cm Second assessment during advanced first stage of labor with a cervix dilation Over 3 cm and less than 10 cm Third assessment during second stage of labor at complete cervix dilation Fourth assessment during the pushing process

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi Slim University Hospital, Tunis, Sidi Daoued La Marsa, Tunisia

REFERENCES:
- [Derived] Dimassi K, Halouani A, Ben Zina F, Khemessi N, Triki A. Regulated Expiratory Methods During Childbirth Process: A Randomized Controlled Trial. J Obstet Gynaecol Can. 2024 Mar;46(3):102265. doi: 10.1016/j.jogc.2023.102265. Epub 2023 Nov 7. PMID 37940044